CLINICAL TRIAL: NCT03624426
Title: Detection and Prevention of Perioperative Nerve Injury Using Automated Somatosensory Evoked Potential Monitoring in Shoulder Arthroplasty Surgery
Brief Title: Detection and Prevention of Nerve Injury in Shoulder Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 108951
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Neuropathy; Nerve Injury
Keywords: nerve monitoring; automated somatosensory evoked potential; nerve injury

STUDY DESIGN:
Intervention Model Description: 1:1 parallel, superiority study
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcome assessor will be blinded. The physicians and operating room nurses, anesthesiologists could not be blinded due to the nature of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated SSEP Monitored Group (Experimental): SSEP monitored group: When a nerve alert is signaled by the automated SSEP device, the surgeon will be informed with the aim to reverse the signal changes. The possible surgical interventions include repositioning the operative arm into a more neutral position, avoidance of excessive traction, removal of retractors, and using a smaller implant to avoid over-correction/traction. The actual intervention will depend on the possible mechanism of nerve injury and treated accordingly.
  Interventions: Device: Automated Somatosensory Evoked Potential device (EPAD@)
- Standard Group (No Intervention): The automated SSEP device will be connected and will be blinded to the surgeon. The screens of the automated SSEP device will be covered by an opaque plastic bag and the alarms will be turned off. No intervention is planned for this group.

INTERVENTIONS:
Device: Automated Somatosensory Evoked Potential device (EPAD@) — After commencement of general anesthesia and during patient positioning, stimulating sensors will be applied to patient wrists and a recording sensor is applied at base of neck posteriorly (at C5 level), forehead and the bilateral wrists. The monitoring will be continued throughout the surgery.
  Arms: Automated SSEP Monitored Group

SUMMARY:
Up to 5% of total shoulder arthroplasty patients experience transient or permanent nerve injury during surgery. In this study, we will monitor the nerve transmission of the patients' arm to detect whether the nerve is functioning normally. This techniques is called somatosensory evoked potential (SSEP) monitoring. In this study, we will assess whether SSEP monitoring could detect nerve abnormalities, alerts the surgical team enabling optimize their surgical intervention and prevent surgical related nerve injury.

DETAILED DESCRIPTION:
Perioperative PNI is a well-recognized but seriously under-investigated complication of general anesthesia. Arguably, such nerve injury may be viewed as being as devastating as spinal cord and cerebral injury, as the resultant functional disabilities may be very comparable.(1) Many such nerve injured patients require prolonged recovery and rehabilitation, while some result in long-term disability and/or litigation due to motor deficits and chronic pain.(2-5) In ASA Closed Claims Analysis PNI was the second most common cause of claims other than death.(6, 7) However, little progress has been made in the past three decades in developing a reliable intraoperative monitoring technique for early detection and prevention. SSEP monitoring is a potential option for preventing PNI. Abnormal SSEP is widely used as a surrogate outcome for PNI in research studies (8-11). Additionally, previous studies (12-17) investigating the use of SSEP for spinal cord or cerebral injury during neurosurgical procedures have incidentally found high incidences of abnormal SSEP (4-7%) due to mal-positioning that was corrected with repositioning; this suggested SSEP could be used to detect intraoperative PNI and that prompt intervention can reverse PNI. However, there have been no further prospective studies to evaluate the diagnostic value of SSEP, or its outcome benefit. This is largely because conventional SSEP is a bulky, expensive and labor-intensive monitoring modality, requiring a technologist for operation and interpretation.(18) Because of these budgetary and logistical limitations, as well as the relative lack of clinical evidence, SSEP is not performed routinely in most surgical centres solely for the purpose of PNI detection. The recent introduction of the Evoked Potential Assessment Device (EPAD®, SafeOp Surgical, Hunt Valley, MD) may be able to overcome these practical barriers. It is a novel, simplified, automated SSEP monitoring device (FDA approved). The key features of EPAD® are its compactness, ease of connectivity via Bluetooth, and its use of surface adhesive electrodes that remove the potential for needle-stick injuries. This device also incorporates an automated progressive signal optimization algorithm, several newly developed artifact rejection and electrocautery suppression technologies as well as an auto-interpretation diagnostic system. It eliminates the need for a designated technician and permits simplified and direct interpretation of the SSEP data for clinicians in the operating room. This device also enables display and storage of raw SSEP data permitting post hoc area-under-curve analysis. (Fig. 3) We have previously evaluated the clinical utility of this automated SSEP device in 33 cardiac surgical patients (19). This pilot study found that automated SSEP monitoring can be performed readily in a busy cardiac operating room. The raw signal quality is reliable and comparable to the conventional SSEP machine. These results indicate that this device is able to eliminate the practical challenges of performing SSEP monitoring and confirmed its feasibility for routine use.(REB# 104826) Surgical-related nerve injury during TSA is one of the highest risk subspecialties leading to postoperative upper limb peripheral neuropathy with reported incidences of 1-4% (20-22). A previous cohort study10, using motor evoked potential and EMG to evaluate the nerve injury during TSA, reported an exceedingly high incidence of intraoperative alerts (56.7% of patients). Importantly, 76.7% (23 of 30) of nerve alerts were reversed with repositioning of the patients' arm and removal of the retractor. Another cohort study11 in shoulder rotator cuff repair reported an even higher incidence of nerve alert (76.5%). Both studies were received Neer research awards from the Orthopedic Society, however neither study has informed the outcome benefit nor has assessed the relationship between cumulative injury, baseline nerve reserve and postoperative neuropathy. Accordingly, we propose to perform single blinded, superiority, parallel design, prospective randomized controlled study to assess the efficacy of the automated SSEP device in preventing PNI during TSA and explore the dose-response relationship of PNI.

ELIGIBILITY:
Inclusion Criteria:

* Adult elective patients undergoing total shoulder arthroplasty surgery using general anesthesia

Exclusion Criteria:

* Patients unable to perform complete neurological examination
* Patients who refuse to participate
* Unable to obtain informed consent.
* Patients who are contraindicated for (or unable to perform) SSEP monitoring
* Patients who have known pre-existing peripheral neuropathy or brachial plexus injury
* Patients who are contraindicated to brachial plexus block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Cumulative duration of abnormal SSEP changes | duration of surgery
  The cumulative duration (min) of abnormal SSEP changes in the operative arm.

SECONDARY OUTCOMES:
New-onset of peripheral neuropathy | 2 weeks, 6 weeks and 3 months
  New-onset peripheral neuropathy of the operative arm at postoperative 6 weeks. A thorough neurologic examination will be performed by an independent assessor before (after brachial plexus catheter inserted), and after the surgery (6 weeks). Any new neurological deficit at postoperative 6 weeks that identified by the independent outcomes assessor will be defined as a positive case.
American shoulder and elbow surgeons standardized shoulder assessment form | 2 weeks, 6 weeks and 3 months
  ASES score is a 100 point scale that consists of two dimensions; pain and daily activity. The pain scale is worth 50 points and the daily activity is worth 50 points. 100 points describes being pain- free and able to complete daily activity with no issues while a score of 0 describes extreme pain and unable to complete daily activities.
Quality of life measure | 2 weeks, 6 weeks and 3 months
  The EQ-5D-5L score consists of two components: a descriptive component to assess five dimensions of quality of life and an EQ visual analogue scale (VAS). The EQ-5D health state index is a single summary index, ranging from 0 to 1 (where 0 denotes death and 1 denotes full health/function), that is weighted to the country/region to describe the five dimensions of EQ-5D.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MBChB, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Wojtkiewicz DM, Saunders J, Domeshek L, Novak CB, Kaskutas V, Mackinnon SE. Social impact of peripheral nerve injuries. Hand (N Y). 2015 Jun;10(2):161-7. doi: 10.1007/s11552-014-9692-0. PMID 26034424
- [Background] Grocott HP, Clark JA, Homi HM, Sharma A. "Other" neurologic complications after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2004 Sep;8(3):213-26. doi: 10.1177/108925320400800304. PMID 15375481
- [Background] Sharma AD, Parmley CL, Sreeram G, Grocott HP. Peripheral nerve injuries during cardiac surgery: risk factors, diagnosis, prognosis, and prevention. Anesth Analg. 2000 Dec;91(6):1358-69. doi: 10.1097/00000539-200012000-00010. No abstract available. PMID 11093980
- [Background] Tajiri O, Tateda T, Sugihara H, Yokoyama H, Nishikido O, Mukumoto C. [Brachial plexus neuropathy following open-heart surgery]. Masui. 2004 Apr;53(4):407-10. Japanese. PMID 15160668
- [Background] Fitzgerald M, McKelvey R. Nerve injury and neuropathic pain - A question of age. Exp Neurol. 2016 Jan;275 Pt 2:296-302. doi: 10.1016/j.expneurol.2015.07.013. Epub 2015 Jul 26. PMID 26220898
- [Background] Kroll DA, Caplan RA, Posner K, Ward RJ, Cheney FW. Nerve injury associated with anesthesia. Anesthesiology. 1990 Aug;73(2):202-7. doi: 10.1097/00000542-199008000-00002. PMID 2382845
- [Background] Cheney FW, Domino KB, Caplan RA, Posner KL. Nerve injury associated with anesthesia: a closed claims analysis. Anesthesiology. 1999 Apr;90(4):1062-9. doi: 10.1097/00000542-199904000-00020. PMID 10201678
- [Background] Jellish WS, Blakeman B, Warf P, Slogoff S. Somatosensory evoked potential monitoring used to compare the effect of three asymmetric sternal retractors on brachial plexus function. Anesth Analg. 1999 Feb;88(2):292-7. doi: 10.1097/00000539-199902000-00012. PMID 9972743
- [Background] Wilent B, Oppenheimer S. Utlility of nerve monitoring during shoulder arthroplasty. Journal of Clinical Neurophysiology 2012; 29 (6): 536
- [Background] Nagda SH, Rogers KJ, Sestokas AK, Getz CL, Ramsey ML, Glaser DL, Williams GR Jr. Neer Award 2005: Peripheral nerve function during shoulder arthroplasty using intraoperative nerve monitoring. J Shoulder Elbow Surg. 2007 May-Jun;16(3 Suppl):S2-8. doi: 10.1016/j.jse.2006.01.016. Epub 2006 Jul 26. PMID 17493556
- [Background] Delaney RA, Freehill MT, Janfaza DR, Vlassakov KV, Higgins LD, Warner JJ. 2014 Neer Award Paper: neuromonitoring the Latarjet procedure. J Shoulder Elbow Surg. 2014 Oct;23(10):1473-80. doi: 10.1016/j.jse.2014.04.003. Epub 2014 Jun 18. PMID 24950948
- [Background] Larson SJ, Gandhoke GS, Kaur J, et al. Incidence of position related neuropraxia in 4489 consecutive patients undergoing spine surgery. Role of SSEP monitoring? Journal of Neurosurgery 2016; 124 (4): A1182
- [Background] Ying T, Wang X, Sun H, Tang Y, Yuan Y, Li S. Clinical Usefulness of Somatosensory Evoked Potentials for Detection of Peripheral Nerve and Brachial Plexus Injury Secondary to Malpositioning in Microvascular Decompression. J Clin Neurophysiol. 2015 Dec;32(6):512-5. doi: 10.1097/WNP.0000000000000212. PMID 26629760
- [Background] Araus-Galdos E, Delgado P, Villalain C, Martin-Velasco V, Castilla JM, Salazar A. Prevention of brachial plexus injury due to positioning of patient in spinal surgery. Value of multimodal intraoperative neuromonitoring (IONM). Clinical Neurophysiology 2011; 122: S113
- [Background] Chung I, Glow JA, Dimopoulos V, Walid MS, Smisson HF, Johnston KW, Robinson JS, Grigorian AA. Upper-limb somatosensory evoked potential monitoring in lumbosacral spine surgery: a prognostic marker for position-related ulnar nerve injury. Spine J. 2009 Apr;9(4):287-95. doi: 10.1016/j.spinee.2008.05.004. Epub 2008 Aug 5. PMID 18684675
- [Background] Labrom RD, Hoskins M, Reilly CW, Tredwell SJ, Wong PK. Clinical usefulness of somatosensory evoked potentials for detection of brachial plexopathy secondary to malpositioning in scoliosis surgery. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2089-93. doi: 10.1097/01.brs.0000179305.89193.46. PMID 16166901
- [Background] Schwartz DM, Drummond DS, Hahn M, Ecker ML, Dormans JP. Prevention of positional brachial plexopathy during surgical correction of scoliosis. J Spinal Disord. 2000 Apr;13(2):178-82. doi: 10.1097/00002517-200004000-00015. PMID 10780696
- [Background] Tamkus A, Rice K. Risk of needle-stick injuries associated with the use of subdermal needle electrodes during intraoperative neurophysiologic monitoring. J Neurosurg Anesthesiol. 2014 Jan;26(1):65-8. doi: 10.1097/ANA.0b013e31829b677c. PMID 23774115
- [Background] Chui J, Murkin JM, Turkstra T, McKenzie N, Guo L, Quantz M. A Novel Automated Somatosensory Evoked Potential (SSEP) Monitoring Device for Detection of Intraoperative Peripheral Nerve Injury in Cardiac Surgery: A Clinical Feasibility Study. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1174-1182. doi: 10.1053/j.jvca.2016.11.024. Epub 2016 Nov 17. PMID 28159523
- [Background] Ladermann A, Lubbeke A, Melis B, Stern R, Christofilopoulos P, Bacle G, Walch G. Prevalence of neurologic lesions after total shoulder arthroplasty. J Bone Joint Surg Am. 2011 Jul 20;93(14):1288-93. doi: 10.2106/JBJS.J.00369. PMID 21792494
- [Background] Carofino BC, Brogan DM, Kircher MF, Elhassan BT, Spinner RJ, Bishop AT, Shin AY. Iatrogenic nerve injuries during shoulder surgery. J Bone Joint Surg Am. 2013 Sep 18;95(18):1667-74. doi: 10.2106/JBJS.L.00238. PMID 24048554
- [Background] Ho E, Cofield RH, Balm MR, Hattrup SJ, Rowland CM. Neurologic complications of surgery for anterior shoulder instability. J Shoulder Elbow Surg. 1999 May-Jun;8(3):266-70. doi: 10.1016/s1058-2746(99)90140-4. PMID 10389084